CLINICAL TRIAL: NCT04465877
Title: Single-blind, Randomized, Placebo-controlled, Multiple Dose Study to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of JTT-662 Administered for 28 Days in Subjects With Type 2 Diabetes Mellitus on Metformin Monotherapy
Brief Title: Study to Evaluate Safety, Tolerability, Pharmacokinetics & Pharmacodynamics of JTT-662 in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akros Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AT662-U-20-003
Record Dates: First submitted 2020-07-01; First posted 2020-07-10 (Actual); Results first posted 2023-01-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: JTT-662; Diabetes; Safety; Tolerability; Pharmacokinetics; Pharmacodynamics
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- JTT-662 5 mg (Experimental): JTT-662 5 mg orally once daily from Day 1 to Day 28, after a single dose of placebo on Day -1
  Interventions: Drug: JTT-662
- JTT-662 10 mg (Experimental): JTT-662 10 mg orally once daily from Day 1 to Day 28, after a single dose of placebo on Day -1
  Interventions: Drug: JTT-662
- JTT-662 20 mg (Experimental): JTT-662 20 mg orally once daily from Day 1 to Day 28, after a single dose of placebo on Day -1
  Interventions: Drug: JTT-662
- Placebo (Placebo Comparator): Placebo orally once daily from Day -1 to Day 28
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JTT-662 — Active drug tablets containing JTT-662
  Arms: JTT-662 10 mg; JTT-662 20 mg; JTT-662 5 mg
Drug: Placebo — Placebo tablets matching in appearance to the active drug tablets
  Arms: Placebo

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of JTT-662 administered once daily for 28 days in subjects with Type 2 diabetes mellitus (T2DM) who are receiving metformin monotherapy

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T2DM for at least 12 weeks prior to the Screening Visit
* Currently treated with a stable oral dose of metformin monotherapy for at least 12 weeks prior to the Screening Visit and until Day -3
* Have a glycosylated hemoglobin (HbA1c) value of between 6.5% and 10.0% at the Screening Visit
* Have a fasting plasma glucose (FPG) value of no more than 280 mg/dL at the Screening Visit and on Day -3
* Body Mass Index (BMI) of 25 to 40 kg/m2 (inclusive)

Exclusion Criteria:

* Known medical history or presence of Type 1 diabetes mellitus, Maturity Onset Diabetes of the Young or secondary forms of diabetes
* Known medical history or presence of diabetic complications
* Have taken anti-diabetic medications (other than metformin) or medications that act mainly in the gastrointestinal tract (e.g., orlistat, acarbose) within 12 weeks prior to the Screening Visit or from the Screening Visit to Day -3
* Have uncontrolled hypertension (systolic blood pressure of at least 160 mmHg or diastolic blood pressure of at least 95 mmHg) at the Screening Visit
* Have impaired renal function (estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-02-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Qps-Mra, Llc, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Written informed consent was obtained prior to performing any study-related procedures. A copy of the informed consent was provided to each subject enrolled in this study. To qualify for the study, subjects were required to satisfy defined criteria.
Pre-assignment Details: Following informed consent signing, screening procedures to confirm eligibility were performed.
  All subjects received a single dose of placebo on Day -1 (Placebo Run-in Period) followed by JTT-662 or placebo once-daily (QD) for 28 consecutive days (Day 1 through Day 28).
Period: Overall Study
Arm/Group | JTT-662 5 mg | JTT-662 10 mg | JTT-662 20 mg | Placebo
Started | 9 | 9 | 10 | 9
Randomized Population (Randomized Population consists of all subjects randomized to receive JTT-662 or placebo on Day 1.) | 9 | 9 | 10 | 9
Safety Population (Safety Population consists of subjects who were randomly assigned to treatment and who received at least one dose of study drug.) | 9 | 9 | 10 | 9
PK (Pharmacokinetic) Population (PK (Pharmacokinetic) Population consists of subjects randomized to JTT-662 treatment groups who received at least one dose of JTT-662 and had available PK data.) | 9 | 9 | 10 | 0
PD (Pharmacodynamic) Population (PD (Pharmacodynamic) Population consists of subjects who were randomly assigned to treatment, received at least one dose of JTT-662 or placebo starting on Day 1 and had evaluable PD data.) | 9 | 9 | 10 | 9
Completed | 9 | 9 | 9 | 9
Not Completed | 0 | 0 | 1 | 0
Not completed — Noncompliant with study requirements | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | JTT-662 5 mg | JTT-662 10 mg | JTT-662 20 mg | Placebo | Total
Number analyzed (Participants) | 9 | 9 | 10 | 9 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 10 | 9 | 35
  >=65 years | 1 | 1 | 0 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 4 | 2 | 16
  Male | 5 | 3 | 6 | 7 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 9 | 10 | 9 | 37
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 1 | 3
  White | 9 | 9 | 8 | 8 | 34
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Treatment-emergent Adverse Events
Description: Treatment-emergent adverse event is defined as any adverse event (untoward medical experience occurring to a subject whether or not it is related to the study drug) with an onset date/time at/after the placebo dosing on Day -1.
Time Frame: 6 Weeks (from Day -1 to the follow-up visit on Day 42)
Population: Safety Population consists of subjects who were randomly assigned to treatment and who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Run-in: Subjects randomized in all 4 treatment groups (JTT-662 5 mg, JTT-662 10 mg, JTT-662 20 mg and Placebo) received a single dose of Placebo on Day -1
Arm/Group | JTT-662 5 mg | JTT-662 10 mg | JTT-662 20 mg | Placebo | Placebo Run-in
Number analyzed (Participants) | 9 | 9 | 10 | 9 | 37
Participants
  Number of subjects with TEAEs | 4 | 7 | 10 | 6 | 3
  Number of subjects with no TEAEs | 5 | 2 | 0 | 3 | 34

2. Primary Outcome: Number of Stools and Type of Stools Based on Bristol Stool Chart
Description: Number of occurrences for each stool type was reported based on their type assessed from Bristol Stool Chart. The Bristol Stool Chart was used to assess the stool shape using a 7-point scale. Where, Type 1 = separate hard lumps, like nuts (hard to pass), Type 2 = sausage-shaped but lumpy, Type 3 = like a sausage but with cracks on the surface, Type 4 = like a sausage or snake, smooth and soft, Type 5 = soft blobs with clear-cut edges (passed easily), Type 6 = fluffy pieces with ragged edges, a mushy stool, Type 7 = watery, no solid pieces; entirely liquid. A score of 1 or 2 indicates constipation while a score of 6 or 7 indicates diarrhea.
Time Frame: 7 Weeks (from Day -6 to the follow-up visit on Day 42)
Population: as for outcome 1
Measure: Number; unit: Number of stools
Arm/Group | JTT-662 5 mg | JTT-662 10 mg | JTT-662 20 mg | Placebo
Number analyzed (Participants) | 9 | 9 | 10 | 9
Number of stools
  Total Number of Stools | 491 | 550 | 815 | 599
  Type 1 | 15 | 3 | 9 | 4
  Type 2 | 31 | 12 | 11 | 17
  Type 3 | 41 | 21 | 18 | 102
  Type 4 | 226 | 173 | 119 | 329
  Type 5 | 63 | 117 | 106 | 97
  Type 6 | 73 | 94 | 242 | 25
  Type 7 | 42 | 130 | 310 | 25

3. Primary Outcome: Trough Concentrations of JTT-662 in Plasma on Days 1, 7, 10, 14, 15, 21 and 28
Description: Trough plasma concentration is the measured concentration at the end of a dosing interval at steady state (taken directly before next administration). Blood samples were collected at specific timepoints to measure trough plasma concentrations of JTT-662 in the subjects randomized to JTT-662 treatment groups.
Time Frame: 28 Days
Population: PK Population consists of subjects randomized to JTT-662 treatment groups who received at least one dose of JTT-662 and had available PK data. The number of subjects on Days 21 and 28 is only 27 since 1 subject in the JTT-662 20 mg group discontinued the study on Day 19.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | JTT-662 5 mg | JTT-662 10 mg | JTT-662 20 mg
Number analyzed (Participants) | 9 | 9 | 10
ng/mL
  Day 1: number analyzed (Participants) | 9 | 8 | 10
  Day 1 | 60.2 (14.4) | 124 (36.0) | 231 (61.9)
  Day 7 | 209 (61.5) | 518 (155) | 845 (359)
  Day 10 | 235 (64.3) | 629 (181) | 959 (449)
  Day 14 | 257 (97.3) | 703 (224) | 1130 (502)
  Day 15: number analyzed (Participants) | 9 | 9 | 9
  Day 15 | 266 (83.7) | 689 (209) | 1140 (475)
  Day 21: number analyzed (Participants) | 9 | 9 | 9
  Day 21 | 281 (100) | 787 (237) | 1180 (665)
  Day 28: number analyzed (Participants) | 9 | 9 | 9
  Day 28 | 292 (103) | 786 (326) | 1190 (583)

4. Primary Outcome: Change From Baseline in AUEC0-4 for Plasma Postprandial Glucose (PPG) Compared to Placebo on Days 1, 14 and 28
Description: Change from baseline in the AUEC0-4 (area under the observed effect-time curve from the start of breakfast until the 4 hour time point) for PPG were calculated using the corresponding Day -1 value as baseline and compared to the placebo values. Negative values represent greater reduction in PPG from baseline values compared to placebo.
Time Frame: Days 1, 14 and 28
Population: PD Population consists of subjects who were randomly assigned to treatment, received at least one dose of JTT-662 or placebo starting on Day 1 and had evaluable PD data. For the JTT-662 20 mg group, number of participants analyzed on Day 28 is 9 since 1 subject did not complete the study.
Measure: Least Squares Mean (90% Confidence Interval); unit: mg*hr/dL
Arm/Group | JTT-662 5 mg | JTT-662 10 mg | JTT-662 20 mg | Placebo
Number analyzed (Participants) | 9 | 9 | 10 | 9
mg*hr/dL
  Day 1 | -0.34 [-55.64 to 54.96] | -98.24 [-153.78 to -42.69] | -88.19 [-140.71 to -35.67] | 1.78 [-54.00 to 57.57]
  Day 14 | -31.22 [-106.31 to 43.88] | -169.40 [-244.67 to -94.13] | -253.57 [-324.85 to -182.29] | -31.55 [-106.99 to 43.89]
  Day 28: number analyzed (Participants) | 9 | 9 | 9 | 9
  Day 28 | -61.17 [-154.63 to 32.28] | -230.87 [-324.46 to -137.28] | -250.64 [-340.71 to -160.58] | -1.83 [-95.55 to 91.90]
Statistical Analysis 1: Comparison: JTT-662 5 mg vs Placebo; Difference between change from baseline in PPG (AUEC0-4) value for JTT-662 5 mg and placebo on Day 1; Test type: Superiority; p = 0.956, Mixed Models Analysis; Mean Difference (Final Values) = -2.12, 95% CI 2-sided [-79.67 to 75.42]
Statistical Analysis 2: Comparison: JTT-662 5 mg vs Placebo; Difference between change from baseline in PPG (AUEC0-4) value for JTT-662 5 mg and placebo on Day 14; Test type: Superiority; p = 0.995, Mixed Models Analysis; Mean Difference (Final Values) = 0.33, 95% CI 2-sided [-105.41 to 106.07]
Statistical Analysis 3: Comparison: JTT-662 5 mg vs Placebo; Difference between change from baseline in PPG (AUEC0-4) value for JTT-662 5 mg and placebo on Day 28; Test type: Superiority; p = 0.366, Mixed Models Analysis; Mean Difference (Final Values) = -59.35, 95% CI 2-sided [-191.15 to 72.45]
Statistical Analysis 4: Comparison: JTT-662 10 mg vs Placebo; Difference between change from baseline in PPG (AUEC0-4) value for JTT-662 10 mg and placebo on Day 1; Test type: Superiority; p = 0.016, Mixed Models Analysis; Mean Difference (Final Values) = -100.02, 95% CI 2-sided [-179.96 to -20.08]
Statistical Analysis 5: Comparison: JTT-662 10 mg vs Placebo; Difference between change from baseline in PPG (AUEC0-4) value for JTT-662 10 mg and placebo on Day 14; Test type: Superiority; p = 0.014, Mixed Models Analysis; Mean Difference (Final Values) = -137.85, 95% CI 2-sided [-245.28 to -30.43]
Statistical Analysis 6: Comparison: JTT-662 10 mg vs Placebo; Difference between change from baseline in PPG (AUEC0-4) value for JTT-662 10 mg and placebo on Day 28; Test type: Superiority; p = 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -229.04, 95% CI 2-sided [-362.17 to -95.91]
Statistical Analysis 7: Comparison: JTT-662 20 mg vs Placebo; Difference between change from baseline in PPG (AUEC0-4) value for JTT-662 20 mg and placebo on Day 1; Test type: Superiority; p = 0.025, Mixed Models Analysis; Mean Difference (Final Values) = -89.98, 95% CI 2-sided [-167.62 to -12.33]
Statistical Analysis 8: Comparison: JTT-662 20 mg vs Placebo; Difference between change from baseline in PPG (AUEC0-4) value for JTT-662 20 mg and placebo on Day 14; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -222.02, 95% CI 2-sided [-326.54 to -117.51]
Statistical Analysis 9: Comparison: JTT-662 20 mg vs Placebo; Difference between change from baseline in PPG (AUEC0-4) value for JTT-662 20 mg and placebo on Day 28; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -248.82, 95% CI 2-sided [-379.35 to -118.28]

ADVERSE EVENTS:
Time Frame: Up to 6 weeks (from Day -1 to the follow-up visit on Day 42)
Description: Safety Population consists of subjects who were randomly assigned to treatment and who received at least one dose of study drug.
Arm/Group | JTT-662 5 mg | JTT-662 10 mg | JTT-662 20 mg | Placebo | Placebo Run-in
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/10 | 0/9 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/10 | 0/9 | 0/37
Other Adverse Events (participants affected / at risk) | 4/9 | 7/9 | 10/10 | 6/9 | 3/37
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | JTT-662 5 mg (N=9) | JTT-662 10 mg (N=9) | JTT-662 20 mg (N=10) | Placebo (N=9) | Placebo Run-in (N=37)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 5 (5) | 10 (12) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications at least 60 days prior to public release. The sponsor will have a review period of 60 days and can embargo communications regarding trial results for an additional period of 60 days from the end of sponsor review period. The sponsor may require removal of any and all confidential information (other than study results) in the communication.

DOCUMENTS (2):
  • Study Protocol (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT04465877/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT04465877/SAP_001.pdf